CLINICAL TRIAL: NCT03514615
Title: A Double Blind, Placebo Controlled, Randomised Dose Escalation Trial to Investigate the Safety and Efficacy of Topical Salbutamol in the Improvement of Scar Appearance When Applied to Approximated Wound Margins in Healthy Volunteers.
Brief Title: A Trial to Assess the Safety and Efficacy of Topical Salbutamol in Healthy Volunteers.
Acronym: SSCART
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: University of Leicester (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 97807
Record Dates: First submitted 2018-02-26; First posted 2018-05-02 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Scarring
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Gel (Placebo Comparator): Each participant will be allocated to only one dosing group. The treatments will be paired anatomically so that for each pair of sites, one closed incision site will receive the active gel and the other placebo.
  Interventions: Procedure: Incision; Drug: Placebo gel
- Active Gel (Experimental): Each participant will be allocated to only one dosing group. The treatments will be paired anatomically so that for each pair of sites, one closed incision site will receive the active gel and the other placebo.
  Interventions: Procedure: Incision; Drug: Active gel

INTERVENTIONS:
Procedure: Incision — A skin incision will be made on the medial aspect of the upper arm.
Drug: Active gel — The incision site on one arm will be dosed with the active gel.
  Arms: Active Gel
Drug: Placebo gel — The incision site on the other arm will be dosed with placebo gel.
  Arms: Placebo Gel

SUMMARY:
This will be a single centre, double-blind, placebo (vehicle) controlled, randomised, dose escalation trial. Three concentrations of topical salbutamol gel will be compared, in a group-wise fashion, with a placebo administration at one incision site on each arm of the trial subjects. Each participant will be allocated to only one dosing group. The treatments will be paired anatomically so that for each pair of sites, one closed incision site will receive the active substance, while the other will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Able, in the opinion of the investigator, and willing to give informed consent
2. Aged 18 - 50 inclusive, with both arms
3. Participants registered on The Over Volunteering Prevention System (TOPS) or equivalent in Leicester.
4. Body mass index within the range 15.0-35.0 kg/m2. Inclusive (i.e. ≥ 15.0 and ≤ 35.0)
5. In the opinion of the investigator, clinically acceptable results for the laboratory tests specified in the trial protocol (see Protocol Section 11.2). All laboratory tests must be performed within 28 days of the subject's first trial dose administration.
6. Women of child bearing potential (WOCBP) must be using a highly effective means of contraception and agree to do so from at least the screening visit until trial end or completion of the trial.

Exclusion Criteria:

1. On direct questioning, have evidence of Left/Right Confusion.
2. On direct questioning and/or physical examination a history or evidence of keloid scarring.
3. On direct questioning have a family history of keloid scarring.
4. Tattoos or previous scars within 3cm of the area to be incised during the trial.
5. Surgery in the area to be incised and have surgical scars within 3cm of this area.
6. History of a bleeding disorder or who are receiving anti-coagulant or anti-platelet therapy.
7. On direct questioning and physical examination, have evidence of any past or present clinically significant disease that may affect the endpoints of the trial. For example: Coagulation disorders, diabetes, immuno-mediated conditions or allergies (including allergic contact dermatitis).
8. Subjects with a clinically significant skin disorder (dermatitis, eczema, psoriasis) that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial.
9. Any clinically significant medical condition or history that would impair wound healing including:

   * Rheumatoid arthritis.
   * Chronic renal impairment for their age.
   * Hepatic impairment (LFTs >3 times upper limit of normal).
   * Congestive heart failure.
   * Pre-existing ischemic heart disease
   * Pulmonary hypertension
   * Hypertrophic obstructive cardiomyopathy
   * Aortic stenosis
   * Current active malignancy or history of malignancy in the last 5 years.
   * Immunosuppression or chemotherapy within the last 12 months.
   * A history of radiotherapy at the areas to be studied.
   * Diabetes mellitus.
   * Subjects with proven diagnosis of thyroid disease
10. A history of hypersensitivity to any of the drugs or dressings used in this trial
11. Currently taking other prescribed treatments:

    * All corticosteroids, whether topically applied or systemic;
    * Any salbutamol containing preparations
    * Other beta-agonists, such as salmeterol
    * Any beta-blockers, such as propranolol
    * Other beta antagonists
    * Adrenaline
12. Undergoing investigations or changes in management for an existing medical condition.
13. History of drug abuse, including cocaine, amphetamines, methamphetamines, opiates or benzodiazepines.
14. In the opinion of the investigator, are unlikely to complete the trial for whatever reason.
15. Any clinically significant neurological impairment or disease, including body dysmorphia.
16. At entry into the trial, any active infection.
17. Pregnant or lactating or planning to become pregnant during the duration of the trial.
18. Not involved with any other clinical trial of medicinal product at the time of consent or 3 months prior.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration | 24 hours
  The primary trial endpoint will be the peak plasma concentration of salbutamol at day 0.

SECONDARY OUTCOMES:
Peak Plasma concentration 2 | 10 days
  The peak plasma concentration of salbutamol at day 10.
Efficacy of treatment using the Global Scar Comparison Scale | 12 months
  Improvement in scar appearance will be assessed using a global appearance scale, referred to as the "Global Scar Comparison Scale" (GSCS), which seeks to assess which one of a pair of scars is visually improved compared to the other. The scale is based on a 200mm Visual Analogue Scale, with "0"mm at the centre indicating no difference between the scars. The extremes of the scale -100mm to +100mm are reserved for one scar becoming imperceptible compared to the other. The assessment will be performed by both the patient and investigator independently at months 7, 9 and 12.
Efficacy of treatment using the Patient Observer Scar Assessment Scale | 12 months
  Improvement in scar appearance will be assessed using the "Patient and Observer Scar Assessment Scale" (POSAS) which is a composite scale made up of sub-scales, that measure 12 items numerically (6 by the patient; scar pain, scar itch, colour differences, scar stiffness, scar thickness and scar irregularity) and six items scored by the investigator (vascularity, pigmentation, thickness, relief, pliability and surface area). The patient sub-scales are scored 1-10 where 1="no, not at all" and 10 = "yes, very much". The clinical sub-scores are also scored 1-10 with 1=normal skin and 10=worst scar imaginable. POSAS is calculated as a total score of all sub-scores. The assessment will be performed by both the patient and investigator independently at months 7, 9 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Johnston, Principal Investigator — University of Leicester
Locations (1):
- Leicester Royal Infirmary, Leicester, United Kingdom